CLINICAL TRIAL: NCT04756141
Title: Continuous Glucose Monitor (CGM) Use in COVID-19 Patients
Brief Title: CGM Use in COVID19 Patients (Infection With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2))
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian G. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-010816
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus; Covid19
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Use (Experimental): Determine CGM accuracy when compared with POC (point of care) glucometers.
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — A CGM will be placed on patients with diabetes mellitus and COVID-19 infection and interstitial glucose will be monitored continuously while the patients are in the hospital.

SUMMARY:
The purpose of this research is to determine if CGM (continuous glucose monitors) used in the hospital in patients with COVID-19 and diabetes treated with insulin will be as accurate as point of care (POC) glucose monitors. Also if found to be accurate, CGM reading data will be used together with POC glucometers to dose insulin therapy.

DETAILED DESCRIPTION:
Study participation involves placement of a continuous glucose monitor (CGM) on the abdomen of hospitalized patients who have a diagnosis of COVID19. The CGM will measure glucose levels every 5 minutes which will be accessible for viewing using a receiver phone placed outside the patient's room and/or an iPad located at the nursing station.

Alarm limits for hypoglycemia and hyperglycemia will be set on the receiver phone for nursing staff to review. These alarms settings will vary depending on whether the patient is on IV insulin infusion vs. subcutaneous (SQ) insulin. The number of glucose checks required with these two types of insulin varies significantly and requires separate handling.

Hospital glucometers will be used to confirm the accuracy of CGM readings during an initial "Adjustment Phase" of the study. If CGMs are found to be accurate, then finger-stick glucometer check frequency will be decreased, and some of the CGM values will be used to dose insulin therapy during the "Utilization Phase" of the study. The instructions for these phases will differ for patients on IV insulin infusion vs. SQ insulin infusion and are detailed in separate protocols. Nursing staff will choose the appropriate protocol at the time of CGM placement based on the type of insulin the patient is receiving.

Different patient variables (demographics, comorbidities, labs and vitals, administered medications) will be collected from electronic health record and will be evaluated to determine if they interfere with CGM readings. At the time of discharge, patients will receive a survey regarding satisfaction with the use of CGM monitors to manage their diabetes during their inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patients with diagnosis of COVID-19 respiratory infection.
* Patient with recent positive SARS-COV2 infection and still positive polymerase chain reaction (PCR) admitted of non-respiratory diagnoses.
* Diagnosis of diabetes mellitus type 1 or type 2.
* Diagnosis of medication (steroid) induced hyperglycemia (persistent glucose more than 180 mg/dl).
* Taking insulin either SQ or IV.

Exclusion Criteria:

* Patient in shock.
* Patient intubated on mechanical ventilation.
* Patient placed on Extracorporeal membrane oxygenation (ECMO).
* Patient taking hydroxyurea.
* Patient taking more than 4g of acetaminophen in 24 hours or more than 1g acetaminophen in 6 hours.
* Pregnant or nursing female patients.
* Patients with skin lesions at the application site that may interfere with placement of the sensor.
* Patients with known allergy to medical grade adhesive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitor (CGM) Use: Continuous Glucose Monitor (CGM): A CGM was placed on patients with diabetes mellitus and COVID-19 infection and interstitial glucose was monitored continuously while the patients were in the hospital.
Period: Overall Study
Arm/Group | Continuous Glucose Monitor (CGM) Use
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Relative Difference (MARD)
Description: Per patient, the absolute relative difference is calculated as the absolute difference between Point of Care (POC) glucose measurements and the nearest Continuous glucose monitor (CGM) measurement (within 5 minutes of POC), divided by the POC glucose value and expressed as a percentage.
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: percentage of MARD
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
percentage of MARD | 10.1 (2.3)

2. Secondary Outcome: CGM Recorded Hypoglycemia Episodes
Description: The total number of hypoglycemia episodes (glucose level below 70 mg/dl).
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Number; unit: hypoglycemia episodes
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
hypoglycemia episodes | 4

3. Secondary Outcome: CGM Recorded Hyperglycemia Episodes
Description: The number of patients that experience GCM recorded hyperglycemia episodes (glucose level above 250 mg/dl).
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
Participants | 19

4. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: MAP is a calculation that checks whether there's enough blood flow to supply blood to all the major organs. Too much resistance and pressure may impede that flow. MAP is the average pressure in the arteries throughout one cardiac cycle. Normal MAP is between 70 and 100 mm Hg
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
mm Hg | 91.8 (12.49)

5. Secondary Outcome: Blood Oxygen Level (SpO2)
Description: SpO2 is a measure of oxygen saturation levels in the blood. It is the percentage of oxygenated hemoglobin (the protein the carries oxygen) compared to the total amount of hemoglobin in the blood. A normal SpO2 level for healthy lungs is typically between 95 and 100 percent.
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: percentage of oxygenated hemoglobin
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
percentage of oxygenated hemoglobin | 94.0 (3.22)

6. Secondary Outcome: CGM Accuracy in Lactic Acidosis.
Description: CGM accuracy via MARD when patients have a lactic acid above 2.2 mmol/L
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Population: Data was not collected nor analyzed
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 0

7. Secondary Outcome: Hospitalization Length of Stay
Description: Total number of days subjects were admitted to the hospital
Time Frame: subject hospital discharge, up to approximately 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
days | 11.0 [4 to 61]

8. Secondary Outcome: Sensor Related Skin Reactions
Description: The number of subjects who experienced sensor related skin reactions
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
Participants | 0

9. Secondary Outcome: Patient Satisfaction Using the Patient Satisfaction Survey
Description: The number of patients who reported being satisfied and very satisfied. The Patient Satisfaction Survey measures the level of patient satisfaction with the question of " How satisfied were you with the nursing staff using a CGM to measure your blood sugar?" the score ranges from 0 (not at all) to 5 (very satisfied).
Time Frame: From date of admission and until discharge from the hospital up to 30 days.
Population: 4 subjects did not complete the survey
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 16
Participants | 12

10. Secondary Outcome: Continuous Glucose Monitor (CGM) Calibrations
Description: The number of calibrations that were performed on the CGM per patient.
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Median (Full Range); unit: calibration per patient
Arm/Group | Continuous Glucose Monitor (CGM) Use
Number analyzed (Participants) | 20
calibration per patient | 2.5 [0 to 25]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 30 days
Arm/Group | Continuous Glucose Monitor (CGM) Use
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Glucose Monitor (CGM) Use (N=20)
Pain (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT04756141/Prot_SAP_000.pdf